CLINICAL TRIAL: NCT03754933
Title: Phase 1/2, Open-label Study Evaluating Safety of Repeat Administration of Ad/PNP-F-araAMP (Ad/PNP Administered Intratumorally Followed by Intravenous Fludarabine Phosphate) in Subjects With Recurrent, Local Head and Neck Cancer
Brief Title: Safety and Efficacy of Repeat Administration of Ad/PNP and Fludarabine Phosphate in Patients With Local Head/Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeoVax, Inc. (Industry)
Collaborators: Stanford University (Other); Emory University (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNP-002; R01FD005746-01A1 (FDA); 14271 (Registry Identifier: IND)
Record Dates: First submitted 2018-10-19; First posted 2018-11-27 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Recurrent Head and Neck Cancer
Keywords: Fludarabine; Adenovirus; Head & neck squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Adenoviridae Infections; Squamous Cell Carcinoma of Head and Neck | interventions — fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ad/PNP + fludarabine phosphate, 5 cycles (Experimental): Ad/PNP + fludarabine phosphate, 5 cycles
  Interventions: Biological: Ad/PNP; Drug: Fludarabine Phosphate

INTERVENTIONS:
Biological: Ad/PNP — Ad/PNP is a replication defective adenoviral vector expressing E. coli Purine Nucleoside Phosphorylase
  Other Names: Gedeptin
Drug: Fludarabine Phosphate — Fludarabine phosphate is an anticancer agent currently used for treatment of patients with chronic lymphocytic leukemia.
  Other Names: Fludara

SUMMARY:
Primary Objective: The primary objective of the study is to evaluate the safety of repeat administration of a dose level of Ad/PNP plus fludarabine phosphate (F-araAMP) which demonstrated anti-tumor activity in patients with advanced head and neck cancer in a completed phase I study.

Secondary Objective: The secondary objective is to evaluate the antitumor activity of repeat administration of Ad/PNP plus F-araAMP.

FDA Office of Orphan Drugs Division is a source of funding for the overall project.

DETAILED DESCRIPTION:
1. Mechanism of action. The study drug, Ad/PNP-F-araAMP (Fludarabine phosphate) consists of a nonreplicating adenoviral vector expressing the E. coli purine nucleoside phosphorylase (PNP) injected intratumorally followed by intravenous administration of F-araAMP. This combination generates 2-fluoroadenine (F-Ade) within the tumor resulting in focal chemotherapeutic activity.

   F-araAMP is an agent that is rapidly cleaved by plasma phosphatases to fludarabine, which is the primary circulating form of the drug and has activity against certain hematological malignancies, but not against solid tumors such as head and neck squamous cell carcinoma (HNSCC). Fludarabine (F-araA) is an adenosine analog and substrate for E. coli PNP, which cleaves the glycosidic bond of F-araA to generate F-Ade. The F-Ade metabolite has shown pronounced activity against human tumor xenografts in mice.

   Many refractory tumors are refractory precisely because they have a very low growth fraction, i.e., a relatively small percentage of tumor cells dividing at any particular point in time. In nonclinical studies, significant in vivo antitumor activity has been demonstrated by F-Ade generation from F-araAMP in tumors in which 2.5 to 10% of cells express the E. coli PNP gene. In addition, anti-tumor effect was seen in patients with advanced solid tumors (melanoma and head and neck cancer) in the higher dose cohorts during a Phase 1 study (see next section).
2. Tumor response with Ad/PNP-F-araAMP in Phase 1 Study. The safety and efficacy of Ad/PNP-F-araAMP has been evaluated in a Phase 1 study, PNP-001 (NCT01310179). Four escalating dose levels were evaluated in 10 subjects with head and neck cancer and 2 subjects with melanoma; clinical activity was observed at the highest dose levels following 3 intratumoral injections of Ad/PNP over 2 days and IV F-araAMP phosphate over 3 days. The overall response rate (CR+PR) was approximately 67% in the 2 highest dose cohorts, Cohorts 3 and 4. Results suggest a dose response effect. The duration of response in the injected tumor was limited, with 4 of 5 responding tumors having disease progression of the injected lesion prior to last follow-up on Day 56, suggesting that repeat administration should be evaluated. Ad/PNP + F-araAMP was well tolerated. No subject experienced a dose-limiting toxicity and none of the subjects discontinued study treatment. Overall, the activity and safety profile of Ad/PNP seen in the Phase 1 study supports further clinical evaluation of repeat administration of Ad/PNP (IT) and F-araAMP phosphate infusion for patients with HNSCC.
3. Purpose of the Study. Based upon the tumor response seen with a single administration of the two highest dose levels of Ad/PNP-F-araAMP in the Phase 1 study (NCT01310179), PNP plans to investigate the safety and assess anti-tumor activity of repeat cycles of injection of Ad/PNP + F-araAMP in patients with advanced head and neck cancer. Subjects in the study will have RECIST 1.1 measurable HNSCC which is amenable to local injection for which there is no effective curative or palliative treatment option. This study population was selected since results from this Phase 1/2 trial are intended to support the safety of repeat dosing in further clinical investigation.
4. Study Design. The trial is designed as a single-arm study to evaluate the safety of repeat cycles of Ad/PNP and F-araAMP in patients with recurrent HNSCC with tumor(s) accessible for injection. Ad/PNP will be injected intratumorally twice on Day 1 and once on Day 2 followed by infusion of F-araAMP daily on Days 3, 4, and 5. Subjects will receive repeat administration of Ad/PNP-F-araAMP every 4 weeks (i.e., each cycle) for 5 cycles or until injected tumor progresses, unacceptable toxicity occurs, no tumor is present for injection, or patient death. Tumor response in the injected tumor(s) will be assessed by physical examination as well as by radiographic imaging. All subjects will be monitored for adverse events during study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Provided Informed Consent
2. Age ≥ 18 years
3. Patients with histologically or cytologically confirmed diagnosis of recurrent cancer of the head and neck region for whom there is no curative treatment option. For the purposes of trial eligibility, cancers of the head and neck shall include, in addition to head and neck squamous cell carcinoma (HNSCC), cutaneous squamous cell primary sites and squamous cell carcinoma of unknown primary presenting with neck lymph nodal disease, as well as nasopharyngeal carcinoma, and salivary gland tumors.
4. All standard or approved treatment options that would provide substantive palliation must have failed, been exhausted, or patient not eligible or willing to use them (for example neuropathy, nephropathy , or hearing loss precluding the use of cisplatin)
5. Tumor mass (primary tumor and/or lymphadenopathy) measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and technically suitable for intratumoral injections (otolaryngologist will determine feasibility). Patients with nodal disease (or metastatic disease) that is needle accessible are eligible. Patients with additional tumors (including distant metastatic disease) beyond the intratumoral injection accessible tumor(s) that are not accessible for intratumoral injection are eligible ONLY if the patient has no other treatment option for the metastatic disease and treatment of local disease may provide the patient some benefit or palliation.
6. Eastern Cooperative Oncology Group performance status of ≤ 2
7. In the judgment of the Investigator, the patient has recovered sufficiently from any previous significant therapy side effects or toxicities prior to Ad/PNP administration.
8. Absolute neutrophil count ≥ 1,500 cells/ul; hemoglobin ≥ 9 g/dl, platelets ≥ 100,000/ul
9. Serum creatinine ≤ 1.5 mg/dl, or calculated creatinine clearance ≥ 60 ml/min
10. Bilirubin ≤ upper limit of normal, alanine aminotransferase ≤ 1.5 x upper limit of normal and/or aspartate aminotransferase ≤ 1.5 x upper limit of normal, alkaline phosphatase ≤ 2.5 x upper limit of normal
11. Prothrombin time (PT)/international normalized ratio (INR) ≤ 1.5 x upper limit of normal
12. Activated partial thromboplastin (aPTT) time ≤ 1.5 x upper limit of normal
13. Female patients must have a negative urine or serum pregnancy at screening (pregnancy test is not required for patients with bilateral oophorectomy and/or hysterectomy or for those patients who are > 1 year postmenopausal)
14. All patients of reproductive potential must agree to use a medically acceptable form of contraception (eg, hormonal birth control, double-barrier method) or abstinence.

Exclusion Criteria:

1. Prior history or current diagnosis of leukemia
2. Have received any gene therapy products or oncolytic viral therapy
3. Receiving allopurinol
4. Received an investigational drug within 30 days prior to first injection of Ad/PNP
5. Received radiation treatment < 4 weeks prior to first injection of Ad/PNP, and does not have any RECIST 1.1 evaluable lesions that are outside the radiation field. (If the patient has RECIST 1.1 evaluable lesions outside the radiation field then they can be included.)
6. Received chemotherapy (systemic anticancer treatment) < 4 weeks prior to first injection of Ad/PNP and has not recovered from all the related side effects. (If the patient has recovered from all related side effects or has reached a new baseline, then they may begin receiving treatment at sooner than 4 weeks)
7. Have significant baseline neuropathy (> Grade 2 based on Common Terminology Criteria for Adverse events [CTCAE] v5.0)
8. Uncontrolled intercurrent disease (e.g., diabetes, hypertension, thyroid disease, active infection)
9. Had within 6 months prior to enrollment: Myocardial infarction, cerebral vascular accident, uncontrolled congestive heart failure, significant liver disease, unstable angina
10. Fever (temperature > 38.1 degrees C orally)
11. Receiving chronic systemic corticosteroids (> 3 weeks) or any chronic immunosuppressive medications within 14 days prior to first injection of Ad/PNP. Subjects receiving short courses of corticosteroids are considered eligible for the study.
12. Receiving anticoagulants other than those to maintain patency of venous lines
13. Women who are pregnant or breast feeding
14. History of HIV infection. No requirement for testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Dimitrios Colevas, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Winship Cancer Institute - Emory University School of Medicine, Atlanta, Georgia
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parker WB, Sorscher EJ. Use of E. coli Purine Nucleoside Phosphorylase in the Treatment of Solid Tumors. Curr Pharm Des. 2017 Nov 8:10.2174/1381612823666171109101851. doi: 10.2174/1381612823666171109101851. Online ahead of print. PMID 29119917
- [Background] Rosenthal EL, Chung TK, Parker WB, Allan PW, Clemons L, Lowman D, Hong J, Hunt FR, Richman J, Conry RM, Mannion K, Carroll WR, Nabell L, Sorscher EJ. Phase I dose-escalating trial of Escherichia coli purine nucleoside phosphorylase and fludarabine gene therapy for advanced solid tumors. Ann Oncol. 2015 Jul;26(7):1481-7. doi: 10.1093/annonc/mdv196. Epub 2015 Apr 21. PMID 25899782

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 subjects provided consent; however, only 8 subjects were assigned to the treatment group as one subject died and one subject was determined ineligible (per protocol entry criteria) prior to treatment assignment.
Period: Overall Study
Arm/Group | Ad/PNP + Fludarabine Phosphate, 5 Cycles
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: lesions
Arm/Group | Ad/PNP + Fludarabine Phosphate, 5 Cycles
Number analyzed (Participants) | 8
Number analyzed (lesions) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Disease History - Duration of Time from Initial Diagnosis (months) [Mean (Standard Deviation); unit: months] — Duration of Time from Initial Diagnosis in months
  months | 44.90 (18.184)
Disease History - Staging at First Diagnosis [Count of Participants; unit: Participants] — Stage 0 - Cancer is only present on the epidermis.
  Stage I - Cancer has grown deep into the skin, but has not spread to nearby lymph nodes or healthy tissues.
  Stage II - Cancer has grown deep into the skin and displays one or more high-risk features (such as metastasis to nerves or lower skin layers), but has not spread to nearby lymph nodes or healthy tissues.
  Stage III - Cancer has grown into lymph nodes, but has not spread to any organs other than the skin.
  Stage IV - Cancer has spread to one or more distant organs, such as the lungs, liver, brain or distant parts of the skin.
  Participants
    II | 1
    III | 3
    IV | 3
    Missing | 1
Disease History - Histological Type [Count of Participants; unit: Participants]
  Squamous cell carcinoma | 6
  Other | 2
Disease History - Progression/Recurrence/Metastasis Specification [Count of Participants; unit: Participants] — Subjects may be counted in more than 1 category
  Participants
    Progression - Local | 1
    Recurrence - Local | 4
    Regional | 1
    Progression - Regional | 3
    Recurrence - Regional | 2
    Metastasis | 5
Disease History - Progression/Recurrence/Metastasis Location [Count of Participants; unit: Participants] — Subjects may be counted in more than one category
  Participants
    Hypopharynx | 1
    Larynx | 1
    Lymph node | 4
    Nasal cavity | 1
    Other | 4
    Pharynx | 2
    Soft tissue | 1
Disease Characteristics at Baseline - Summary of Diameters of Target Lesions [Mean (Standard Deviation); unit: mm] — Tumor mass (primary tumor and/or lymphadenopathy) must have been technically suitable for intratumoral injections (as determined by otolaryngologist). Subjects with nodal disease (or metastatic disease) that were needle accessible were eligible. Subjects with additional tumors (including distant metastatic disease) beyond the intratumoral injection accessible tumor(s) that were not accessible for intratumoral injection were eligible ONLY if the subject had no other treatment option for the metastatic disease and treatment of local disease might provide the subject some benefit or palliation.
  mm | 92.93 (76.255)
Disease Characteristics at Baseline - Summary of Diameters of For-Injection Lesions [Mean (Standard Deviation); unit: mm] — Tumor mass (primary tumor and/or lymphadenopathy) must have been technically suitable for intratumoral injections (as determined by otolaryngologist). Subjects with nodal disease (or metastatic disease) that were needle accessible were eligible. Subjects with additional tumors (including distant metastatic disease) beyond the intratumoral injection accessible tumor(s) that were not accessible for intratumoral injection were eligible ONLY if the subject had no other treatment option for the metastatic disease and treatment of local disease might provide the subject some benefit or palliation.
  mm | 50.30 (36.542)
Disease Characteristics at Baseline - ECOG [Count of Participants; unit: Participants] — Grade 0: Fully active, able to carry out all normal activities without restriction; considered the best performance status.
  Grade 1: Restricted in strenuous activity but still ambulatory and able to perform light work.
  Grade 2: Able to perform all self-care activities but unable to work, up and about for more than 50% of waking hours.
  Participants
    Grade 0 | 1
    Grade 1 | 5
    Grade 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety Measures (Adverse Events and Laboratory Parameters) With Repeat Cycles of Treatment.
Description: Safety measures evaluated by medical history, physical examination, vital signs, inspection of tumor site, performance status, EKG, chest X-ray (CXR), blood chemistry, hematology, CD4/CD8 T-cell counts, urinalysis, PT/PTT, blood sample for adenovirus, urine for adenovirus, F-Ade plasma level, blood sample for antibody against adenovirus, and monitoring adverse events.
Time Frame: up to 7 months
Population: Defined as all participants who received any intratumoral administrations of Ad/PNP or any infusion of F-araAMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad/PNP + Fludarabine Phosphate, 5 Cycles
Number analyzed (Participants) | 8
Participants
  Serious Adverse Events | 5
  Fatal SAEs | 0
  Any TEAE | 8
  Any TEAE Related to Study Treatment | 8
  Any TEAE Related to Non-Study Treatment | 1
  Any TEAE Grade 3 or Greater | 7
  Dose Limiting Toxicity TEAE | 0
  Any TEAE Leading to Study Discontinuation | 1
  Any TEAE Grade 3 or Greater Related to Study Treatment | 3
  Any Serious TEAE | 5

2. Secondary Outcome: Best Overall Response for Injected Tumors During 5 Cycles of Treatment as Determined by RECIST 1.1.
Description: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: up to 7 months
Population: All participants who received at least three intratumoral administrations of Ad/PNP and any infusion of F-araAMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Ad/PNP + Fludarabine Phosphate, 5 Cycles
Number analyzed (Participants) | 8
Participants
  Stable Disease | 3
  Progressive Disease | 2
  Not Evaluable | 3

3. Secondary Outcome: Progression Free Survival (PFS) - Time From First Intratumoral Injection to Date of Progression or Death, Calculated in Months
Description: Time to Event (Progression or Death) was defined as time from first intratumoral injection to date of progression or death for any cause, whichever occurred first, and was calculated, in months, as: (Date of first PD (Progressive Disease) or death or censoring - date of first intratumoral injection + 1) / 30.4375. PD was defined, based on the protocol-defined criteria for response in For-Injection tumors, as at least a 20% increase in the longest diameter (LD) of the injected lesions, taking as reference the smallest LD recorded on study (this includes the baseline LD if that is the smallest on study; note: appearance of one or more new lesions was considered progression in assessing overall tumor response.). PFS derivation did not include tumor assessments collected after the end of study treatment as these were not planned for collection beyond the final cycle.
Time Frame: up to 7 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ad/PNP + Fludarabine Phosphate, 5 Cycles
Number analyzed (Participants) | 8
Months | 7.0 [.39 to NA] — Not enough participants achieved response to calculate upper 95% CI

4. Secondary Outcome: Probability of No Progressive Disease or Death and 95% CI Up to 6 Months (%)
Description: Time to PD or death was defined as time from the first intratumoral injection to date of progression or death for any cause, whichever occurs first, and was calculated, in months, as: (Date of first PD or death or censoring - date of first intratumoral injection + 1) / 30.4375.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Ad/PNP + Fludarabine Phosphate, 5 Cycles
Number analyzed (Participants) | 8
percentage of subjects | 56.3 [14.7 to 84.2]

5. Secondary Outcome: Overall Survival (OS) - Time From First Intratumoral Injection to Date of Death up to 60 Days Post Last Injection
Description: Time to death was defined as time from the first intratumoral injection to date of death for any cause, and was calculated, in months, as: (Date of death or censoring - date of the first intratumoral injection + 1) / 30.4375. Subjects still alive as of the data cut-off date were censored on the last known alive date from mortality status follow up. For subjects that were lost to follow up, the last visit in the database or last contact date where the subject was documented to be alive was used to estimate last known date alive.
Time Frame: up to 7 months
Population: All participants who received at least three intratumoral administrations of Ad/PNP and any infusion of F-araAMP.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ad/PNP + Fludarabine Phosphate, 5 Cycles
Number analyzed (Participants) | 8
Months | 7.0 [.69 to NA] — Not enough participants achieved response to calculate upper 95% CI

6. Secondary Outcome: Probability of No Death and 95% CI up to 1 Month and up to 6 Months
Description: Time to death was defined as time from the first intratumoral injection to date of death for any cause, and was calculated, in months, as: Date of death or censoring - date of the first intratumoral injection + 1 / 30.4375.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Ad/PNP + Fludarabine Phosphate, 5 Cycles
Number analyzed (Participants) | 8
percentage of subjects
  Up to 1 month | 87.5 [38.7 to 98.1]
  Up to 6 months | 72.9 [27.6 to 92.5]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from signing of informed consent up to 6 months. Serious and Other Adverse Events were assessed from initiation of study treatment (Day 1) up to 6 months.
Description: All adverse events regardless of seriousness or relationship to study drug were recorded. Only All-Cause Mortality was assessed in the 2 participants that were enrolled but not randomized. All-Cause mortality, SAEs and Other Adverse Events were assessed in the safety population, which was defined as all participants who received any intratumoral administrations of Ad/PNP or an infusion of F-araAMP.
Groups:
- Participants Who Were Enrolled But Not Randomized: Participants who were enrolled but not randomized
Arm/Group | Ad/PNP + Fludarabine Phosphate, 5 Cycles | Participants Who Were Enrolled But Not Randomized
All-Cause Mortality (participants affected / at risk) | 3/8 | 1/2
Serious Adverse Events (participants affected / at risk) | 5/8 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ad/PNP + Fludarabine Phosphate, 5 Cycles (N=8) | Participants Who Were Enrolled But Not Randomized (N=0)
Pneumonia (Infections and infestations) | 1 (1) | NA — Pneumonia
Fever (General disorders) | 1 (1) | NA — Fever
Vomiting (Gastrointestinal disorders) | 1 (1) | NA — Vomiting
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | NA — Supraventricular tachycardia
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA — Tumor hemorrhage
Dysphagia (Gastrointestinal disorders) | 1 (1) | NA — Dysphagia
Dehydration (Metabolism and nutrition disorders) | 1 (1) | NA — Dehydration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ad/PNP + Fludarabine Phosphate, 5 Cycles (N=8) | Participants Who Were Enrolled But Not Randomized (N=0)
Injection Site Pain (General disorders) | 6 (12) | NA
Fatigue (General disorders) | 4 (4) | NA
Injection Site Bruising (General disorders) | 2 (3) | NA
Pyrexia (General disorders) | 1 (1) | NA
Chest Pain (General disorders) | 1 (1) | NA
Chills (General disorders) | 1 (1) | NA
Injection Site Oedma (General disorders) | 1 (1) | NA
Localized Oedema (General disorders) | 1 (1) | NA
Non-Cardiac Chest Pain (General disorders) | 1 (1) | NA
Oedema (General disorders) | 1 (1) | NA
Pain (General disorders) | 1 (1) | NA
Swelling Face (General disorders) | 1 (1) | NA
Nausea (Gastrointestinal disorders) | 4 (5) | NA
Dysphagia (Gastrointestinal disorders) | 4 (5) | NA
Vomiting (Gastrointestinal disorders) | 1 (2) | NA
Constipation (Gastrointestinal disorders) | 1 (1) | NA
Dry Mouth (Gastrointestinal disorders) | 1 (1) | NA
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | NA
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Tumor Hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | NA
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Hypertension (Vascular disorders) | 4 (5) | NA
Hypotension (Vascular disorders) | 1 (2) | NA
Infestation (Infections and infestations) | 1 (1) | NA
Wound Infection (Infections and infestations) | 1 (1) | NA
Decreased Appetite (Metabolism and nutrition disorders) | 2 (3) | NA
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 1 (1) | NA
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | NA
Dizziness (Nervous system disorders) | 1 (1) | NA
Headache (Nervous system disorders) | 1 (2) | NA
Somnolence (Nervous system disorders) | 1 (1) | NA
Tachycardia (Cardiac disorders) | 1 (1) | NA
Lymphocyte Count Decreased (Investigations) | 1 (1) | NA
Weight Decreased (Investigations) | 1 (1) | NA
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Anemia (Blood and lymphatic system disorders) | 1 (1) | NA
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | NA
Ocular Hyperaemia (Eye disorders) | 1 (1) | NA
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | NA
Insomnia (Psychiatric disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that a MULTI CENTER PUBLICATION (MCP) coordinated by SPONSOR will be the first publication to present the pooled STUDY results. PI agrees not to independently publish, present or otherwise disclose any results of the STUDY until a MCP is published. Following the MCP, or if the MCP is not submitted for publication within18 months of database lock or any earlier termination of the STUDY, PI shall have the right to publish or present materials related to the STUDY.

DOCUMENTS (2):
  • Study Protocol (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT03754933/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT03754933/SAP_001.pdf